CLINICAL TRIAL: NCT03647917
Title: A Pilot, Randomized, Single-Blind, Controlled Study Evaluating the Use of Platelet Rich Plasma (PRP) and Microneedling for Facial and Hand Skin Rejuvenation
Brief Title: A Pilot Study on the Use of Platelet Rich Plasma (PRP) for Facial and Hand Skin Rejuvenation
Acronym: PRP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alison J. Bruce, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 17-005431
Record Dates: First submitted 2018-06-29; First posted 2018-08-27 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Skin Aging of Face and Hands

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Plasma, Left face and hands (Experimental): Subjects will receive PRP on left half of face and saline solution on right half of face through injections via filler injection technique followed by microneedling, and will also receive PRP on dorsal part of left hand and saline solution on dorsal part of right hand through injections via filler injection technique. Microneedling will not be performed on the hands.
  Injections will take place every 4 weeks for a total of 3 treatments.
  Interventions: Biological: Platelet Rich Plasma
- Platelet Rich Plasma, Right face and hands (Experimental): Subjects will receive PRP on right half of face and saline solution on left half of face through injections via filler injection technique followed by microneedling, and will also receive PRP on dorsal part of right hand and saline solution on dorsal part of left hand, through injections via filler injection technique. Microneedling will not be performed on the hands.
  Injections will take place every 4 weeks for a total of 3 treatments.
  Interventions: Biological: Platelet Rich Plasma

INTERVENTIONS:
Biological: Platelet Rich Plasma — Autologous Platelet Rich Plasma (PRP) will be isolated from the blood collected from each subject at each treatment time point.
  Face: Using a 30 gage needle, about four points of PRP or saline will be injected into the malar area; about six points will be injected into the mandibular area; and seven points will be injected into the forehead (0.2 mL per point) with a total volume of approximately 3.5 mL. PRP and saline application will be followed by microneedling.
  Hands: Using a 30 gage needle about 1 cc of PRP or saline will be injected into the dorsal area of the hands (0.2mL per point) at five points. No microneedling will be performed on the hands.
  Arms: Platelet Rich Plasma, Left face and hands
Biological: Platelet Rich Plasma — Autologous Platelet Rich Plasma (PRP) will be isolated from the blood collected from each subject at each treatment time point.
  Face: Using a 30 gage needle, about four points of PRP or saline will be injected into the malar area; about six points will be injected into the mandibular area; and seven points will be injected into the forehead (0.2 mL per point) with a total volume of approximately 3.5 mL. PRP and saline application will be followed by microneedling.
  Hands: Using a 30 gage needle about 1 cc of PRP or saline will be injected into the dorsal area of the hands (0.2mL per point) at five points. No microneedling will be performed on the hands.
  Arms: Platelet Rich Plasma, Right face and hands

SUMMARY:
The overall goal of this study is to develop regenerative cell therapy for use in female patients with aging skin. The primary objective of this proposal is to conduct a pilot study on the efficacy and safety of using PRP to treat this condition in females.

DETAILED DESCRIPTION:
Recently, there has been interest in treatments which are orientated to more biologically regenerative therapies, with several studies demonstrating successful use for PRP in skin rejuvenation. Although PRP is widely used in clinical dermatology, experimental studies confirming the effects of PRP on aged fibroblasts are very limited.

PRP contains concentrated platelet cells derived from autologous whole blood that are believed to induce the synthesis of collagen and other matrix components by stimulating the activation of fibroblasts, thus rejuvenating the skin when injected into an area of collagen degeneration. In this proposal we will examine whether PRP therapy provides similar or better rejuvenating capacity in women compared to saline solution. The study will be a randomized, controlled trial comparing microneedling with PRP to microneedling with saline solution, in females aged 45 and over with skin aging of face. This study will also compare PRP to saline (given through injections via filler injection technique) in females with aging skin of the hands. Microneedling will not be performed on the hands.

ELIGIBILITY:
Inclusion Criteria

1. Only female patients are eligible
2. Patients must be 45 years of age or older
3. Patients must have signs of skin aging on face (wrinkles, rough texture, skin atrophy and skin laxity) and hands (loss of fat tissue and visibility of veins and tendons).
4. Patients must have been on stable birth control for the past 6 months if able to conceive
5. Patients are able and willing to provide written informed consent after the study is fully explained

Exclusion Criteria

1. Patients with clinically abnormal platelet count, serum chemistry, or screening laboratory results as reviewed by the Principal Investigator
2. Patients who have had any cosmetic procedures meant to address skin aging of face and hands 3 months prior to enrollment
3. Patients who have had resurfacing laser on face or hands within one year prior to enrollment
4. Patients taking anti-rheumatic disease medication (including methotrexate or other anti-metabolites) within the 3 months prior to study entry
5. Patients who are pregnant or currently breast-feeding
6. Patients with systemic, rheumatic, or inflammatory disease or who are immunosuppressed
7. Patients with ongoing infectious disease, including HIV and hepatitis
8. Patients with history of significant cardiovascular, renal, hepatic, endocrine disease, cancer, or diabetes
9. Patients participating in a study of an experimental drug or medical device within 30 days of study entry
10. Patients with history of platelet disorders, bone marrow aplasia, sepsis, or cancer
11. Patients taking anti-aggregating therapy
12. Patients on anticoagulant therapy
13. Patients with history of keloid formation
14. Patients with uncontrolled diabetes
15. Patients with active skin disease or skin infection on the intended treatment areas, at baseline

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Wrinkle Severity Rating Scale (WSRS) | 24 weeks
  The Wrinkle Severity Rating Scale assesses the presence and severity of wrinkles at rest in a rating scale from 0 to 4, where 0 means no visible wrinkles, 1 means minimal wrinkles, 2 means shallow wrinkles, 3 means moderately deep wrinkles and 4 means very deep wrinkles.

SECONDARY OUTCOMES:
Hand Grading Scale | 24 weeks
  The Hand Grading Scale assesses signs of hand aging based on loss of fat tissue and visibility of veins and tendons. It is rating scale form 0 to 4 where 0 means no loss of fat tissue, 1 means mild loss of fat tissue and slight visibility of veins, 2 means moderate loss of fat tissue and mild visibility of veins and tendons, 3 means severe loss of fat tissue and moderate visibility of veins and tendons and 4 means very severe loss of fat tissue and marked visibility of veins and tendons.

CONTACTS AND LOCATIONS:
Overall Officials: Alison J Bruce, MD, Principal Investigator — Mayo Clinic; Thais P Pincelli, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials